CLINICAL TRIAL: NCT04516980
Title: Cross-cultural Translation, Adaptation and Psychometric Validation of the Functional Ankle Instability (IdFAI) in an Italian Population With or Without Ankle Instability - A Non-interventional Web-based Cross-sectional Study
Brief Title: Validation of the Identification of Functional Ankle Instability (IdFAI) in Italian
Acronym: IdFAI-I
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Other Study IDs: IdFAI-I
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Ankle Sprains
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with ankle sprain.: Participants with ankle sprain
  Interventions: Other: Questionnaires administration
- Participants without ankle sprain: Participants without ankle sprain
  Interventions: Other: Questionnaires administration

INTERVENTIONS:
Other: Questionnaires administration — Administration of Identification of Functional Ankle Instability (IdFAI) and the following assessment scales: Self-reported question assess the ankle instability as functional/stable or not functional/unstable, Foot and Ankle ability Measure Italian Version - Activity Daily Living (FAAM-I/ADL), Short-form 36-item Health Survey Italian Version (SF-36), Numeric Rate Scale pain (NRS Pain), Visual Analogic Scale Ankle Instability (VAS ankle instability).
  After a week the participants will fill in the following questionnaires: Identification of Functional Ankle Instability (IdFAI), Numeric Rate Scale pain (NRS Pain), Visual Analogic Scale Ankle Instability (Vas ankle instability) with the additional question to measure the change in complaints.

SUMMARY:
The purpose of the study is actually the translation, cultural adaptation and psychometric validation in the Italian Version of the Identification of Functional Ankle Instability (IdFAI) English Version for use in outpatient clinics in non-English subjects to objectify chronic ankle instability.

DETAILED DESCRIPTION:
The hypothesis is to translate and culturally adapt the scale successfully and demonstrate a good factorial structure and psychometric properties, replicating the results of the original English version of the questionnaire

ELIGIBILITY:
Participants without ankle sprain.

1. Age ≥ 18aa
2. Speak Italian on a daily basis
3. No pathologies or surgical treatments in the lower limbs currently or in the past

Participants with ankle sprain.

Inclusion Criteria

1. Age ≥ 18aa
2. Speak Italian on a daily basis
3. At least one ankle sprain
4. Recurrent sprain to the same ankle and/or sensation of ankle instability and/or 'giving way'

Exclusion Criteria

1. Inability to understand written Italian
2. Acute lower extremity injury occurred in the three months preceding the compilation of the questionnaire
3. History of others lower extremity musculoskeletal diseases or injuries of other joints (i.e, hip, knee), previous ankle fractures or systemic pathologies (i.e., neurological disorders, rheumatoid arthritis) currently or in the past
4. History of surgical treatments in either lower limb (bones, joints, nerves)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects, speaking Italian, without lower limbs current disease or history of lower limbs disease or surgical tretmens in the lower limbs.
  Adult subjects, speaking Italian, with at least one ankle sprain and recurrent sprain to the same ankle and/or sensation of ankle instability and/or 'giving way'
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Psychometric parameter 1 validation of the IdFAI scale. | One week
  Sample Size homogeneity
Psychometric parameter 2 validation of the IdFAI scale. | One week
  Discriminant validity
Psychometric parameter 3 validation of the IdFAI scale. | One week
  Internal consistency
Psychometric parameter 4 validation of the IdFAI scale. | One week
  Construct validity
Psychometric parameter 5 validation of the IdFAI scale. | One week
  Test-retest reliability
Psychometric parameter 6 validation of the IdFAI scale. | One week
  Criterion validity: convergent and divergent validity
Psychometric parameter 7 validation of the IdFAI scale. | One week
  Floor and ceiling effects

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Martinato, PhD, Study Director — University of Padova

IPD SHARING:
Plan to Share IPD: Undecided